CLINICAL TRIAL: NCT06968559
Title: Effect of Early Dexamethasone on Major Complications and All-cause Mortality in Severe Burns
Acronym: DEXA-BURN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC24_0442; 2024-517708-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Severe Burns
MeSH Terms: conditions — Burns | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 0.2 mg/kg of ideal body weight (IBW) IV (at a maximum of 20 mg per day) will be blindly infused from day 1 to day 5
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo: one IV administration per day from day 1 to day 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 0.2 mg/kg of ideal body weight (IBW) IV (at a maximum of 20 mg per day) will be blindly infused from day 1 to day 5;
  Arms: Dexamethasone
Drug: Placebo — Placebo: one IV administration per day from day 1 to day 5.
  Arms: Placebo

SUMMARY:
Burns affect more than 11 million people worldwide each year. These injuries are responsible for severe morbidity resulting in a high societal burden and account for more than 180,000 yearly deaths especially in low- and middle-income countries.

Major burns induce an important local and systemic inflammatory response that may be overwhelmed. This inflammation is a physiological phenomenon that favours the healing of tissues. However, the overproduction of inflammatory mediators might lead to an exacerbated Systemic Inflammatory Response Syndrome (SIRS). Recently the total body surface area (TBSA) burned has shown to be well correlated to persistent elevation of pro-inflammatory mediators (such as IL-6). This SIRS, in turn, contributes to the enhanced risk of sepsis, acute respiratory distress syndromes (ARDS) and organ failures in general such as acute kidney injuries (AKI), most of those occurring within the first week of admission.

Corticosteroids (CS) have already proven their effectiveness against SIRS-induced organ dysfunction or mortality in acute medicine notably in septic shock, polytraumatized patients and more recently in the treatment of viral or non-viral ARDS without increasing the risk of secondary bacterial complications or significant side effects . Indeed the recent SCCM Guidelines clearly advocate for the use of CS in severe community-acquired pneumonia, septic shock and ARDS. The investigators recently performed a large multicenter, double-blinded randomized controlled trial (the PACMAN trial, PHRC-N 2016) including 1222 patients scheduled for major surgery in which the investigators observed a major decrease in CRP blood concentrations in the dexamethasone arm. The rate of AKI and the need for mechanical ventilation were also significantly reduced in the intervention arm. ICU Patients with severe burns undergo several surgeries, including major procedures (excision, skin grafts), rendering them quite similar to those in the PACMAN trial in terms of inflammatory response. Very few side effects (hyperglycemia mainly) easily overcome in ICU are usually reported with the use of low-to-moderate dose of CS.

In severe burn patients, very few data are available to date, two retrospective case control studies and a small prospective randomized trial showed promising results when using CS but high quality evidence is lacking.

The investigators hypothesise here that the use of dexamethasone after major burns, the prototypic model of inflammatory response in surgical ICU patients, would limit SIRS-induced organ failure and/or all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ Age ≤ 80 years old.
* Total burn surface area ≥ 20%, measured by a trained expert upon admission
* Invasive mechanical ventilation at the time of inclusion
* Within 48 hours of the burn injury
* Informed and signed written consent of the next-of-kin, legal representative (trusteeship, guardianship) or emergency procedure in the absence of a legal representative.
* Affiliation with French social security system or beneficiary from such system

Exclusion Criteria:

* Imminent death and a do-not-resuscitate order

  * Medical history of hypersensitivity to dexamethasone and hypersensitivity to all of its excipients
  * Pregnancy (attested by a pregnancy test for women of childbearing age) and/or breastfeeding women
  * Participation to another interventional study involving a drug with known interactions with dexamethasone
  * Uncontrolled viral hepatitis or invasive fungal infection at the time of inclusion
  * Prolonged administration of steroids in the last 90 days (>0.3 mg/kg/day of equivalent prednisolone)
  * Moderate-to-severe ARDS upon admission (according to Berlin definition criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2029-02-07 (Estimated); Study Completion 2029-02-07 (Estimated)

PRIMARY OUTCOMES:
Major complications | 28 days
  It's a hierarchic procedure. Major complications defined as moderate to severe ARDS (using Berlin definition criteria) or AKI KDIGO 2 to 3 within 28 days
All-cause mortality at day 90 | 90 days

SECONDARY OUTCOMES:
Hospital-acquired infections | 28 days
  Hospital-acquired pneumonia (using the joint definition from the Infectious Diseases Society of America and American Thoracic Society) within 28 days
Hospital-acquired infections | 28 days
  Catheter-related bloodstream infections within 28 daysDiseases Society of America and American Thoracic Society) within 28 days
Hospital-acquired infections | 28 days
  other infections, including skin infections (diagnosis confirmed by an independent adjudication committee) with or without bacteraemia within 28 days
Hospital-acquired infections | 28 days
  Antibiotic-free days on day 28
Respiratory complications | 28 days
  ARDS (using Berlin Criteria definition) on day 28
Respiratory complications | 28 days
  Invasive ventilator-free days on day 28
ICU Length-of-Stay | 28 days
  ICU Length-of-Stay
Hospital Length-of-Stay | 28 days
  Hospital Length-of-Stay
risks of organ dysfunction | 14 days
  SOFA scores
risks of organ dysfunction | 28 days
  KDIGO stages 2 and 3 AKI
General tolerance of the treatment | 28 days
  Number of Participants with Hyperglycemia
specific tolerance of the treatment on skin lesions | 28 days
  surgical site infections confirmed by an independent adjudication committee,
Timing of first surgery | 28 days
  Timing of first surgery on the main endpoint
Impact of treatment on serum CRP Levels | 14 days
  Serum CRP levels on day 0, day 1, day 3, day 7 and day 14
General tolerance of the treatment | 28 days
  Number of Participants with hypernatremia
General tolerance of the treatment | 28 days
  Number of Participants with hypokalaemia
General tolerance of the treatment | 28 days
  Number of Participants with gastrointestinal bleeding
General tolerance of the treatment | 28 days
  Number of Participants with acquired-weakness

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Tours, Chambray-lès-Tours
  - CHU Lille, Lille
  - CHU de Lyon, Lyon
  - Aphm Hopital La Timone, Marseille
  - CHR Metz, Metz
  - CHU Montpellier, Montpellier
  - Chu Nantes, Nantes
  - HU Saint-Louis Lariboisière, Paris
  - CHU Bordeaux, Pessac
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No